CLINICAL TRIAL: NCT05079945
Title: Tractography and Diffusion Tensor Imaging of the Human Spinal Cord in Healthy Subjects : Anatomical Atlas
Acronym: TRACTOCORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL21_0265; 2021-A02277-34 (Other: N°ID-RCB)
Record Dates: First submitted 2021-09-21; First posted 2021-10-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer
Keywords: Tractography, DTI, MRI, spinal cord

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spinal cord Tractography (Experimental): Healthy volunteer having the tractography exam
  Interventions: Procedure: Spinal cord Tractography in order to differentiate spinal tracts.

INTERVENTIONS:
Procedure: Spinal cord Tractography in order to differentiate spinal tracts. — Spinal cord tractography using DTI MRI sequences of the brain and spinal cord, in order to differentiate tracts at the spinal cord level; and by performing a stitching process between Brain and Spinal cord DTI sequences.

SUMMARY:
Today, Spinal cord pathologies, whether are tumoral, vascular, traumatic, malformative, inflammatory, or degenerative still constitute a major medico-surgical challenge due to the particular anatomy of the spinal cord. Indeed, the spinal fibers (whether they have a sensory or motor function) are all condensed in an extremely small volume. To date, there is no reliable technique to know the precise position of the spinal tracts specifically involved in the sensory and motor functions of the upper and lower limbs.

The purpose of this study is to evaluate the feasibility for differentiating spinal tracts by tractography from a cerebral Diffusion tensor imaging (DTI) Magnetic Resonance Imaging (MRI) sequence (associated with an anatomical sequence) by performing a stitching process with spinal cord DTI MRI sequence, in healthy subjects. The criterion of differentiation of the tracts will be assessed by highlighting already known cerebral tracts (cortico-spinal fibers, spinothalamic, posterior cord) and which will be monitored at the spinal level.

ELIGIBILITY:
Inclusion Criteria:

* patient> 18 years old
* Healthy volunteer
* Social insured in France
* Patient who signed the informed consent of the study

Exclusion Criteria:

* Medical or surgical history of disease that may affect the central nervous system, or the spine
* History of spine or spinal cord trauma.
* Spinal osteoarthritis which can lead to a medullary hyper signal.
* Contraindication to MRI: claustrophobia, pace-maker, defibrillator, metallic foreign bodies, etc.
* Subjects benefiting from legal protection (curatorship, guardianship or safeguard of justice).
* Pregnant and / or breastfeeding woman.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Spinal tracts differentiation and identification | date of Tractography procedure (DTI MRI)
  Percentage of complete tracts identified among healthy volunteer

SECONDARY OUTCOMES:
Spinal cord Tracts Atlas | 12 months (end of recruitment and exams)
  Elaboration of a tracts classification using a algorithm based on the type, the volume and the fraction of anisotropy and mean diffusivity of each tract

CONTACTS AND LOCATIONS:
Overall Officials: DAULEAC Corentin, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Dauleac Corentin, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dauleac C, Mertens P, Frindel C, Jacquesson T, Cotton F. Atlas-guided brain projection tracts: From regions of interest to tractography 3D rendering. J Anat. 2025 May;246(5):732-744. doi: 10.1111/joa.14120. Epub 2024 Aug 11. PMID 39129322